CLINICAL TRIAL: NCT04885452
Title: Prevention of COVID-19 Complications in High-risk Subjects Infected by SARS-CoV-2 and Eligible for Treatment Under a Cohort ATU ('Autorisation Temporaire d'Utilisation') or or Authorisation for Early Access (AAP). A Prospective Cohort.
Brief Title: Prevention of COVID-19 Complications in High-risk Subjects Infected by SARS-CoV-2 and Eligible for Treatment Under a Cohort ATU ('Autorisation Temporaire d'Utilisation') OR or Authorisation for Early Access (AAP). A Prospectvie Cohort.
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS0003S COCOPREV
Record Dates: First submitted 2021-05-05; First posted 2021-05-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV Infection; Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients treated with casirivimab/imdevimab according to the ATU protocol
  Interventions: Other: biobank
- Patients treated with bamlanivimab/etesevimab according to the ATU protocol
  Interventions: Other: biobank
- Patients treated with Xevudy according to the authorisation for early access (AAP) protocol
  Interventions: Other: biobank
- Patients treated with Paxlovid according to the authorisation for early access (AAP) protocol
  Interventions: Other: biobank

INTERVENTIONS:
Other: biobank — * Blood samples (biobank) at Day 0, Day 7, Month 1 and possibly Month 3 (only for the first 100 participants) (serum, plasma and whole blood)
  * For participants in the immunological ancillary study: additional blood sampling at Day 0, Day 7 and Month 1 (PBMC)
  * Nasopharyngeal swabs: Day 0, Day 7 (Day 14 and Day 21 if RT-PCR positive respectively at Day 7 and Day 14)
  * Specific nasopharyngeal swabs in hospitalized patients: Day 3, Day 5

SUMMARY:
This is a prospective, multicentric, non comparative study aiming to evaluate the clinical and virological evolution of high-risk patients infected with SARS-CoV-2 treated withtin the framework of a cohort ATU ('Autorisation temporaire d'utilisation') or authorisation for early access (AAP) delivered by the French drug agency (ANSM).

ELIGIBILITY:
Inclusion Criteria:

* Adults with the criteria for COVID-19 treatment within the French compassionate program (ATU/AAP)
* Adults covered by the French social health coverage
* Adults who signed the informed consent form

Exclusion Criteria:

* Exclusion criteria described in the French compassionate program (ATU/AAP)
* Patient participating in another biomedical research with an exclusion period ongoing at inclusion
* Vulnerable patient (adults legally protected: under judicial protection, guardianship, or supervision, persons deprived of their liberty)
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with SARS-CoV-2 referred by their doctor (general practitioner, specialist, SOS doctor, etc.) to a prescribing center authorized to prescribe and deliver treatments benefiting from an ATU/AAP.
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients hospitalized (if the patient was outpatient) or whose hospitalization was extended for complications from COVID-19 within 1 month of symtoms' onset. | Month 1

SECONDARY OUTCOMES:
Percentage of patients hospitalized whatever the reason | Month 1 and 3
Percentage of patients with an WHO score >= 5 | Month 1
Percentage of patients staying in an Intensive Care Unit in the month following symptoms' onset | Month 1
Percentage of patients who died from COVID-19 complications and any other reason | Month 1
Percentage of patients presenting a adverse event and percentage of treatment discontinuation caused by those adverse events | Month 1
Time between first symptoms and treatment and the reasons for this delay | Day 0
Virological response | Day 7 for ambulatory patients, Day 3, 5 and 7 for hospitalized patients
  Percentage of virological response defined by CT>=31 or negative PCR test +
Virological criteria linked to the emergence of resistance | from inclusion until a negative PCR test or Ct ≥31 is obtained
  Percentage of patients included developing resistance variants, genotypic and phenotypic characterization of resistance variants
Percentage of patients with positive anti-N and anti-S serology | Day 0 and Month 3
anti-S antibody level | Day 0 and Month 3
Flow cytometry cartography of myeloid response | Day 0, 7 and Month 1
  Flow cytometry cartography of myeloid (functional subtypes of monocytes and dendritic cells) response
Flow cytometry cartography of T-lymphocyte response | Day 0, 7 and Month 1
  Flow cytometry cartography of T-lymphocyte (conventional T-lymphocytes by identifying naïve, memory and effector Th1, Th2, Tfh and Th17 T-lymphocytes, NK and gamma-delta T-lymphocytes, regulatory T-lymphocytes; surface and intracellular markers) response
Flow cytometry cartography of B-lymphocyte response | Day 0, 7 and Month 1
  Flow cytometry cartography of B-lymphocyte (transitional, naïve, memory T-lymphocyte with or without isotypic switching, plasmablasts) response
Dosing of a wide range of cytokines and chemokines (IFNalpha, IFNgamma, IL-6, IL-1, IL-8, IL-15, IL-18, IL1-RA, IL-7, IL-10, CXCL10, CXCL13, CCL2 and CCL3) using the Meso Scale Discovery approach | Day 0, 7 and Month 1
Clinical and biological predictors (clinical parameters, treatment received, virological criteria (cycle threshold (CT), variants) of the onset of complications from COVID19, hospitalization, death | from inclusion until the end of the follow-up (Month 1 or Month 3)
  Identication of clinical and biological predictors of the onset of complications from COVID19, hospitalization, death by a logistic model or survival model (RMST): the response variable is the occurrence of a complication, hospitalization, death or the average survival at 1 month on these different criteria; the covariates are the parameters at inclusion, the treatment received, the virological criteria (CT, variants) which can be considered as a time-dependent covariate
Clinical and biological predictive factors (clinical parameters, treatment received, virological criteria (cycle threshold (CT), variants)) linked to the neutralizing serological response: non-response, duration of the response | from inclusion until the end of the follow-up (Month 1 or Month 3)
  Identification of clinical and biological predictive factors (clinical parameters, treatment received, virological criteria (cycle threshold (CT), variants)) linked to the neutralizing serological response: non-response, duration of the response by a logistic model or mixed model for repeated measures
Clinical and biological predictors (clinical parameters, treatment received, virological criteria) of viral response (viral genotypes, emergence of resistant strains) | from inclusion until the end of the follow-up (Month 1 or Month 3)
  Identification of clinical and biological predictive factors related to the virological response (viral genotypes, emergence of resistant strains) by a logistic model: the response variable is RT-PCR negativation at D7 (or CT≥31), the covariates are the parameters at inclusion, the treatment received, the virological criteria at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Youri Yordanov, Dr, Principal Investigator — Saint Antoine Hospital
Locations (37):
- France (37):
  - CH Agen-Nerac, Agen
  - CHU d'Angers, Angers
  - CHR Metz-Thionville, Ars-Laquenexy
  - Hôpital Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien - Hématologie, Corbeil-Essonnes
  - Centre Hospitalier Sud Francilien - Néphrologie, Corbeil-Essonnes
  - CHU de Dijon, Dijon
  - CHU de Martinique, Fort-de-France
  - Hôpital Bicêtre - Médecine interne, Le Kremlin-Bicêtre
  - Hôpital Bicêtre - SMIT, Le Kremlin-Bicêtre
  - CHU de Limoges, Limoges
  - Hospices Civils de Lyon (HCL), Lyon
  - CHU de Montpellier, Montpellier
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - Hôpital Lariboisière - SMIT, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Bichat Claude-Bernard, Paris
  - Hôpital Tenon, Paris
  - Hôpital Bichat Claude-Bernard - SAU, Paris
  - Hôpital Lariboisière - SAU SMUR, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Saint Antoine - SAU, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Hôpitaux Cochin - Port Royal, Paris
  - CHI Poissy St Germain en Laye, Poissy
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CH de Tarbes, Tarbes
  - CHU de Toulouse - IUCT - Oncopole, Toulouse
  - CHU de Toulouse, Toulouse
  - CH de Tourcoing, Tourcoing
  - CHRU de Tours - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruel T, Vrignaud LL, Porrot F, Staropoli I, Planas D, Guivel-Benhassine F, Puech J, Prot M, Munier S, Henry-Bolland W, Soulie C, Zafilaza K, Lusivika-Nzinga C, Meledge ML, Dorival C, Molino D, Pere H, Yordanov Y, Simon-Loriere E, Veyer D, Carrat F, Schwartz O, Marcelin AG, Martin-Blondel G; ANRS 0003S CoCoPrev Study Group. Antiviral activities of sotrovimab against BQ.1.1 and XBB.1.5 in sera of treated patients. medRxiv [Preprint]. 2023 May 30:2023.05.25.23290512. doi: 10.1101/2023.05.25.23290512. PMID 37398037
- [Background] Bruel T, Vrignaud LL, Porrot F, Staropoli I, Planas D, Guivel-Benhassine F, Puech J, Prot M, Munier S, Bolland WH, Soulie C, Zafilaza K, Lusivika-Nzinga C, Meledge ML, Dorival C, Molino D, Pere H, Yordanov Y, Simon-Loriere E, Veyer D, Carrat F, Schwartz O, Marcelin AG, Martin-Blondel G; ANRS 0003S CoCoPrev Study Group. Sotrovimab therapy elicits antiviral activities against Omicron BQ.1.1 and XBB.1.5 in sera of immunocompromised patients. Med. 2023 Oct 13;4(10):664-667. doi: 10.1016/j.medj.2023.07.007. PMID 37837962
- [Background] Martin-Blondel G, Marcelin AG, Soulie C, Kaisaridi S, Lusivika-Nzinga C, Zafilaza K, Dorival C, Nailler L, Boston A, Ronchetti AM, Melenotte C, Cabie A, Choquet C, Trinh-Duc A, Lacombe K, Gaube G, Coustilleres F, Pourcher V, Martellosio JP, Peiffer-Smadja N, Chauveau M, Housset P, Piroth L, Devaux M, Pialoux G, Martin A, Dubee V, Frey J, Le Bot A, Cazanave C, Petua P, Liblau R, Carrat F, Yordanov Y. Time to negative PCR conversion amongst high-risk patients with mild-to-moderate Omicron BA.1 and BA.2 COVID-19 treated with sotrovimab or nirmatrelvir. Clin Microbiol Infect. 2023 Apr;29(4):543.e5-543.e9. doi: 10.1016/j.cmi.2022.12.016. Epub 2022 Dec 28. PMID 36586513
- [Background] Martin-Blondel G, Marcelin AG, Soulie C, Kaisaridi S, Lusivika-Nzinga C, Dorival C, Nailler L, Boston A, Melenotte C, Gaube G, Choquet C, Liblau R, Carrat F, Yordanov Y; COCOPREV Study Group. Outcome of very high-risk patients treated by Sotrovimab for mild-to-moderate COVID-19 Omicron, a prospective cohort study (the ANRS 0003S COCOPREV study). J Infect. 2022 Jun;84(6):e101-e104. doi: 10.1016/j.jinf.2022.04.010. Epub 2022 Apr 7. No abstract available. PMID 35398409